CLINICAL TRIAL: NCT03753022
Title: Effects of PEEP on Parameters of Tissue Perfusion and Clinical Outcomes After Coronary Artery Bypass Graft Surgery - a Randomized Clinical Trial
Brief Title: Effects of PEEP on Parameters of Tissue Perfusion in Patients Post Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Vanessa Marques Ferreira (Unknown)
Responsible Party: Principal Investigator, Solange Guizilini, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 89704818.6.0000.5505
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting; Acute Lung Injury
Keywords: Acute Lung Injury; postoperative of cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease; Acute Lung Injury

STUDY DESIGN:
Intervention Model Description: The study was planned in 3 groups. Group G5 (control group: no changes will be made to the value of PEEP). Group G10 [after 30 minutes of admission (time 0) the PEEP will be raised to 10 cmH2O (time1) for 30 minutes and then returned to 5 cm H2O (time 2)]. Group G15 [after 30 minutes of admission (time 0) the PEEP will be raised to 15 cmH2O (time 1) for 30 minutes and then returned to 5 cm H2O (time 2)].
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group G5 (Sham Comparator): Patients submitted to CABG and peep 5
  Interventions: Other: Group G5
- Group G10 (Experimental): Patients submitted to CABG and peep 10
  Interventions: Other: Group G10
- Group G15 (Experimental): Patients submitted to CABG and peep 15
  Interventions: Other: Group G15

INTERVENTIONS:
Other: Group G5 — Submitted to peep 5
  Arms: Group G5
Other: Group G10 — Submitted to peep 10
  Arms: Group G10
Other: Group G15 — Submitted to peep 15
  Arms: Group G15

SUMMARY:
Pulmonary dysfunction is a condition inherent in cardiac surgery because of various interventions, such as general anesthesia, a median sternotomy, cardiopulmonary bypass and establishment of internal thoracic artery dissection.

In situations when there is a deterioration in oxygenation, increased positive pressure on the airways end pressure (PEEP) can be used as therapeutic mode by reversing severe hypoxemia resulting pulmonary shunt. But the use of PEEP has been associated to reduced cardiac output, due mainly to decrease systemic venous return consequent to increased intrathoracic pressure, and thus might reduce tissue oxygenation. Moreover, the increased transpulmonary gradient may also impair right ventricular ejection exacerbating the hemodynamic consequences in some patients, which in clinical practice this diagnosis may be difficult to perform.

In hypovolemic patients or those with cardiac changes may become even more pronounced, resulting in accentuation of low flow and systemic hypotension entailing changes in markers of tissue perfusion commonly measured by venous saturation central difference venoarterial carbon dioxide and lactate. The hypothesis of the investigators is that PEEP of 10 cmH2O and 15 cmH2O can be applied to reverse lung damage in patients in the immediate postoperative myocardial revascularization without repercussion tissue importantly in markers of tissue perfusion.

The objective is to evaluate the effects of different optimization levels of PEEP on gas exchange and influences the tissue perfusion after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized study and will be performed on patients who accept coronary artery bypass grafting with cardiopulmonary bypass, the conscious openness to participate in the study. Age, sex, body mass index (BMI), smoking habits, diagnosis, additional diseases, drugs used, surgery, intervention, peroperative supportive treatments, left ventricular ejection fraction, post operative blood and cardiopulmonary bypass (CPB) time (min), cross clamp time (min), duration of operation, postoperative extubation period, intensive care day of hospitalization, day of hospitalization will be recorded.The study was planned in 3 groups. Group G5 (control group: no changes will be made to the value of PEEP). Group G10 [after 30 minutes of admission (time 0) the PEEP will be raised to 10 cmH2O (time1) for 30 minutes and then returned to 5 cmH2O (time 2)]. Group G15 [after 30 minutes of admission (time 0) the PEEP will be raised to 15 cmH2O (time 1) for 30 minutes and then returned to 5 cm H2O (time 2)]. At each time of protocol (0, 1 and 2) will be collected: arterial blood gas measurements (partial pressure of arterial oxygen [PaO2] and partial pressure of carbon dioxide ([PaCO2]), the ratio between the partial oxygen pressure, inspired oxygen fraction (PaO2/FiO2) and pH. Also, will be performed parameters of tissue perfusion: central venous oxygen saturation ([SVO2]), arterial blood lactate, venoarterial CO2 difference ([Dif VA CO2]) and vital signs. In all other respects, treatment will follow the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* elective and isolated CABG, ejection fraction greater than 40%

Exclusion Criteria:

* patients with a diagnosis of pulmonary disease, emergency surgery and mechanical ventilation prior to surgery.

Postoperative patients who had radiological abnormalities suggestive of pneumothorax, atrial or ventricular arrhythmias, electrical ischemic changes on ECG, pulse pressure variation of more than 13, hemodynamic instability characterized by mean arterial pressure less than 60 mmHg, nor epinephrine greater than 0.5 mcg/Kg/ min and the presence of increased bleeding through the drains (greater than 2 ml \ kg \ h) the protocol was discontinued and the patient excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary events | Through study completion, an average of 24 hours after surgery
  Pleural effusion was considered relevant when exceeding the phrenicocostal angle and fluid drainage was monitored hourly. Atelectasis was acknowledged when a clear atelectasis radiologic shadow exceeded 15 mm in width, with linear atelectasis
Arterial oxygenation | Immediately after arrival at the intensive care unit until the end of protocol (around 5 hours)
  arterial blood gas measurements (partial pressure of arterial oxygen [PaO2]
Tissue oxygenation | Immediately after arrival at the intensive care unit until the end of protocol (around 5 hours)
  (central venous oxygen saturation , arterial blood lactate and venoarterial CO2 difference

SECONDARY OUTCOMES:
Length of intensive care unit (ICU) stay | From the day of surgery up to ICU discharge, maximum censoring at day 28 after surgery ]
  Days since surgery until ICU discharge
Length of Hospital Stay | From the day of surgery up to Hospital discharge, maximum censoring at day 28 after surgery ]
  Days since surgery until Hospital discharge
Duration of mechanical ventilation | Through study completion, an average of 24 hours after surgery
  Hours since surgery until extubation

IPD SHARING:
Plan to Share IPD: Undecided